CLINICAL TRIAL: NCT00482261
Title: Phase II Trial of Low Dose Lenalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma (Rev-Lite) in Patients at High Risk for Myelosuppression
Brief Title: A Study of Low Dose Lenalidomide and Dexamethasone in Relapsed/Refractory Myeloma in Patients at High Risk for Myelosuppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-PI-0103; 07/04
Record Dates: First submitted 2007-06-03; First posted 2007-06-05 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: myeloma; relapse; refractory; elderly; lenalidomide
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — Lenalidomide; Dexamethasone; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- len-dex (Experimental): Drug: Lenalidomide 15mg daily, days 1-21 of a 28 day cycle for 4 cycles. Patients who get stable disease or better will then receive 15mg on days 1-21 from cycle 5 onwards; Drug: dexamethasone 20mg day 1-4, 9-12, 17-20 for 4 cycles. Patients who get stable disease or better will then get dexamethasone 20mg on days 1-4 of a 28 day cycle, from cycle 5 onwards
  Interventions: Drug: Lenalidomide; Drug: dexamethasone; Drug: aspirin

INTERVENTIONS:
Drug: Lenalidomide — 15mg daily, days 1-21 of a 28 day cycle for 4 cycles. Patients who get stable disease or better will then receive 15mg on days 1-21 from cycle 5 onwards
Drug: dexamethasone — 20mg day 1-4, 9-12, 17-20 for 4 cycles. Patients who get stable disease or better will then get dexamethasone 20mg on days 1-4 of a 28 day cycle, from cycle 5 onwards
Drug: aspirin — 100mg/day

SUMMARY:
The purpose of this study is to see whether combination of low dose lenalidomide(10mg)+ dexamethasone is equally effective in treating relapsed/refractory myeloma in the group of elderly patients and other patients at risk of myelosuppression, whilst producing less side effects, especially myelosuppression compared to the higher dose of lenalidomide of 25mg used in the MM-009 and MM-010 trials.

DETAILED DESCRIPTION:
Lenalidomide has proven efficacy in myeloma. In the Phase I studies with lenalidomide monotherapy, responses were observed at doses of 5mg, 10mg and 25mg. The dose limiting toxicity of lenalidomide monotherapy was myelosuppression·

In the International MM-010 and MM-009 studies, lenalidomide was administered at 25mg d1-d21 (with pulse dexamethasone) of a 28 day cycle. Although the overall response rate and time to progression were impressive, a significant toxicity was myelosuppression. The average age in these 2 studies was approximately 63 years, some 7 years lower than the median age for myeloma. The median number of prior therapies was 2. Thus, if lenalidomide therapy is to be optimally applied in an older and/or more heavily pre-treated population, a simpler, less toxic regimen would be valuable. Low dose (15mg) lenalidomide (Rev-Lite) with dexamethasone may achieve this goal·

Based on analysis of the MM009 and MM010 data the patients at highest risk for myelosuppression and subsequent dose reduction were those over the age of 60 years (approx 30% risk which increased to approx 50% by 70 years).It is hypothesized that patients with lower base-line platelets may also be at higher risk of lenalidomide-induced myelosuppression. Little is known about lenalidomide tolerance in patients with impaired renal function, consequently patients with relatively poorer renal function will also be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign consent form.
2. Must meet one of following age group requirements at the time of signing consent form.

   1. age 18-59 years
   2. >59 years
3. Patients 18-59 years are eligible only if:

   * platelets between 50-74x109/L or
   * calculated GFR between 20ml/min and 59ml/min
4. Able to adhere to the study visit schedule and other protocol requirements.
5. Subject was previously diagnosed with multiple myeloma based on standard diagnostic criteria.
6. Must have relapsed or refractory disease.
7. Measurable disease, defined as follows:

   * For secretory multiple myeloma: measurable disease is defined as any quantifiable serum monoclonal protein value (generally, but not necessarily, >5g/L of M-Protein). If the M band is <5g/L, then the serum free light chains(SFLC) must be assessed and if >100mg/L will also be used to measure disease response. Where applicable, urine light-chain excretion of ≥200 mg/24 hours will also be used to measure disease response.
   * For light chain disease (M band in serum <5g/L but measurable FLC in urine): measurable disease is defined by either urine FLC OR the presence of serum FLC (must be >100mg/L). Investigators can use either test (or both) but must use the same method throughout the trial.
   * For non-secretory multiple myeloma (no M-protein in serum or urine by immunofixation): measurable disease is defined by soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan).
8. Patient has a life-expectancy ≥3 months.
9. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
10. ECOG performance status of ≤2 at study entry
11. Laboratory test results within these ranges:

    * Absolute neutrophil count ³ 1.0 x 109/L (can be supported with growth factor)
    * Total bilirubin ≤1.5 mg/dL
    * AST (SGOT) or ALT (SGPT) ≤2 x UL
12. For females subjects:

    * Must have two negative pregnancy tests (sensitivity ≥ 50 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug.
    * Females of childbearing potential (FCBP)† must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.
13. Male Subjects:

    * Must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
    * Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure.
14. Disease free of prior malignancies for ≥3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
15. Able to take aspirin daily as prophylactic anticoagulation. (patients intolerant to ASA may use low molecular weight heparin).

Exclusion Criteria:

1. Dexamethasone resistant myeloma based on last therapy. Patients are defined as being refractory to high-dose dexamethasone if they achieved less than a partial response, or developed progressive disease within 6 months of discontinuing dexamethasone, or dexamethasone was discontinued because of ≥Grade 3 dexamethasone-related toxicity. High-dose dexamethasone therapy is defined as >500mg dexamethasone or equivalent over a 10-week period, whether administered alone or as part of the VAD regimen.
2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
3. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
5. Use of any other experimental drug or therapy within 28 days of baseline.
6. Known hypersensitivity to thalidomide.
7. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
8. Any prior use of lenalidomide.
9. Concurrent use of other anti-cancer agents or treatments.
10. Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
Time To Progression | 2 years
Duration of Response | 2 years
Safety and toxicity | continuous
Prognostic factors associated with ORR, TTP, OS | 2 years
Compare OTT, TTP an toxicities to MM-009/MM-010 data | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miles H Prince, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Cooke RE, Gherardin NA, Harrison SJ, Quach H, Godfrey DI, Prince M, Koldej R, Ritchie DS. Spontaneous onset and transplant models of the Vk*MYC mouse show immunological sequelae comparable to human multiple myeloma. J Transl Med. 2016 Sep 6;14(1):259. doi: 10.1186/s12967-016-0994-6. PMID 27599546